CLINICAL TRIAL: NCT01613014
Title: A Phase 2, Double-Blind, Randomized, Placebo Controlled Trial to Assess the Efficacy of ABT-436 for Alcohol Dependence
Brief Title: ABT-436 for Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCIG-004
Record Dates: First submitted 2012-06-04; First posted 2012-06-06 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Alcohol Dependence; Alcohol Abuse; Alcohol Use Disorders; Alcoholism
Keywords: Alcohol; Alcohol Dependence; Alcohol Abuse; Alcohol Use Disorders; Alcoholism
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar Pill (Placebo Comparator): Matched Placebo sugar pill - target dose 2 pills BID
  Interventions: Drug: Matched Placebo - Sugar Pill
- ABT-436 (Active Comparator): ABT-436 Target dose of 400 mg BID
  Interventions: Drug: ABT-436

INTERVENTIONS:
Drug: ABT-436 — Target dose - 400mg BID
  Arms: ABT-436
Drug: Matched Placebo - Sugar Pill — Target Dose - 2 pills BID
  Arms: Sugar Pill

SUMMARY:
The primary efficacy endpoint examines the hypothesis that ABT-436 will decrease the weekly percentage of heavy drinking days during Study Weeks 2 through 12 (Days 8-84) as compared to placebo. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.

DETAILED DESCRIPTION:
Adrenocorticotropic hormone (ACTH) release from the pituitary gland via V1B stimulation is central to the hypothalamus-pituitary-adrenal (HPA) axis stress response (Carrasco & Van de Kar-2003, Herman & Cullinan-1997, Sapolsky et al-2000; Tsigos & Chrousos-2002). Chronic dysregulation of the HPA axis is common in major depressive disorder, anxiety disorders, and substance abuse disorders characterized by elevated AVP, increased responsiveness to AVP, as well as either increased or decreased overall HPA axis activity or responsiveness (Dinan & Scott-2005). HPA axis normalization via pituitary V1B antagonism is a mechanism for potential ABT-436 efficacy in these disorders (Schüle et al-2009). Limbic V1B antagonism in the brain may also contribute to efficacy (Roper et al-2011).

Alcohol dependence, or alcoholism, is characterized by a chronic relapsing course, in which alcohol-associated cues and stress are known relapse triggers (Brownell et al-1986, Heilig & Egli-2006, Sinha & Li-2007). Recent research suggests that neural systems mediating behavioral stress responses may offer useful targets for pharmacotherapy of alcoholism. In animal models, excessive alcohol consumption that results from a history of alcohol dependence is accompanied by increased behavioral sensitivity to stress (Heilig & Koob-2007). Preclinical studies have shown that V1B antagonists can attenuate reinstatement of heroin and alcohol self-administration, and block dependence-induced exaggeration of alcohol intake, in rats. V1B antagonists have also been shown to block stress-induced reinstatement of drug and alcohol seeking in ethanol dependent rats (Zhou-2011). For these reasons the NIAAA Clinical Investigations Group (NCIG) proposes to test ABT-436 in a Phase 2, proof of concept trial for the treatment of alcohol dependence.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age and no more than 65 years of age.
* Have a current (past 12 months) DSM-IV-TR diagnosis of alcohol dependence.
* Be seeking treatment for alcohol dependence and desire a reduction or cessation of drinking.

Exclusion Criteria:

* current (past 12 months) abuse or dependence on any psychoactive substance other than alcohol, caffeine and nicotine, including sedatives and hypnotics, as defined by DSM-IV-TR criteria.
* positive urine toxicology screen performed during screening or baseline.
* been hospitalized for alcohol intoxication delirium, alcohol withdrawal delirium, alcohol-induced persisting dementia or amnestic disorder, or have had an alcohol withdrawal seizure, alcohol-induced psychotic disorder with a primary diagnosis of alcohol dependence or a history of any seizure disorder.
* Have any of the following, based on DSM-IV-TR criteria as assessed using the MINI:

  1. Current, past, or lifetime diagnosis of psychotic disorders (note schizophrenia is diagnosed under the psychotic disorder module of the MINI)
  2. Current or past diagnosis of bipolar disorder,
  3. Current or past year major depressive episode,
  4. Current (past 3 months) eating disorder (anorexia or bulimia), or
  5. Current (within past year) diagnosis of panic disorder with or without agoraphobia,
  6. Anti-social personality disorder.
* Have any underlying medical condition that could exacerbate during trial participation causing hospitalization, surgery, and/or the need to use exclusionary medications to treat condition.
* Be pregnant or breast-feeding or have plans to become pregnant at any time during the study.
* Have a clinically significant abnormal laboratory value;
* Hemoglobin A1c value > 7%.
* Have a clinically significant ECG as determined by the investigator or abnormal ECG heart rate (<45 or > 100 bpm or QTc interval corrected for heart rate using the Fridericia formula (QTcF) > 450 msec.
* Have HIV or Hepatitis A, B or C.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-02; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raye Litten, PhD, Principal Investigator — National Institute on Alcohol Abuse and Alcoholism (NIAAA)
Locations (5):
- United States (5):
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Boston Medical Center, Quincy, Massachusetts
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sugar Pill | ABT-436
Started | 75 | 75
Completed | 57 | 63
Not Completed | 18 | 12

BASELINE CHARACTERISTICS:
Population: 144 represents the modified intention to treat population (mITT) - took at least one dose of medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | ABT-436 | Total
Number analyzed (Participants) | 71 | 73 | 144
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 71 | 73 | 144
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (11.6) | 45.8 (10.2) | 45.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 27 | 52
  Male | 46 | 46 | 92
Region of Enrollment [Number; unit: participants]
  United States | 71 | 73 | 144

OUTCOME MEASURES:

1. Primary Outcome: Weekly Percentage of Heaving Drinking Days
Description: The primary objective of this study is to assess the efficacy of ABT-436 to reduce the weekly percentage of heavy drinking days (reduction in drinking) in subjects with alcohol dependence confirmed by DSM-IV-TR criteria. A "heavy drinking day" is 4 or more drinks per drinking day for women and 5 or more drinks per drinking day for men.
  The outcome measure was averaged across weeks 2-12.
Time Frame: Weeks 2-12
Population: Models are based on a mITT population that included subjects who received at least one dose of medication (N=144; ABT-436=73, placebo=71). One additional placebo subject had no drinking data during the maintenance period, and one ABT-436 subject was missing data on a baseline covariate, resulting in an analyzable N=142 (ABT-436=72, placebo=70).
Measure: Least Squares Mean (95% Confidence Interval); unit: weekly percentage of heavy drinking days
Arm/Group | Sugar Pill | ABT-436
Number analyzed (Participants) | 70 | 72
weekly percentage of heavy drinking days | 37.6 [29.2 to 45.9] | 31.3 [23.4 to 39.2]

ADVERSE EVENTS:
Description: The sample size for the adverse event table is 144 which is the mITT population - subjects who took at least one dose of medication.
Arm/Group | Sugar Pill | ABT-436
Serious Adverse Events (participants affected / at risk) | 1/71 | 2/73
Other Adverse Events (participants affected / at risk) | 67/71 | 73/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sugar Pill (N=71) | ABT-436 (N=73)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) — From a bee sting
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Peptic Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sugar Pill (N=71) | ABT-436 (N=73)
Diarrhoea (Gastrointestinal disorders) | 14 | 37
Headache (Nervous system disorders) | 18 | 17
Nausea (Gastrointestinal disorders) | 9 | 18
Nasopharyngitis (Gastrointestinal disorders) | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 8 | 5
Blood Creatine Phosphokinase (Blood and lymphatic system disorders) | 6 | 7
Vomiting (Gastrointestinal disorders) | 5 | 7
Dizziness (Nervous system disorders) | 4 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 3 | 7
Dyspepsia (Gastrointestinal disorders) | 4 | 5
Irritability (General disorders) | 4 | 5
Eosinophil Count increased (Investigations) | 3 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Disorientation (Psychiatric disorders) | 4 | 4
Abdominal Distension (Gastrointestinal disorders) | 2 | 5
Abdominal Pain (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 4 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Rash (Skin and subcutaneous tissue disorders) | 4 | 3
Flatulence (Gastrointestinal disorders) | 2 | 4
Rhinitis (Infections and infestations) | 1 | 5
Neutrophil Count Increased (Immune system disorders) | 4 | 2
Red blood cells urine positive (Investigations) | 2 | 4
Anxiety (Psychiatric disorders) | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 1
Asthenia (General disorders) | 0 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No